CLINICAL TRIAL: NCT00172991
Title: Adiponectin Gene and Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9100208420
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2003-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Genetic studies of coronary artery disease, restenosis after angioplasty or stenting, focusing on renin-angiotensin system genes and adiponectin gene, and their interactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving angiography

Exclusion Criteria:

* Patients receiving angioplasty and reluctant for the study

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ti Tsai, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan